CLINICAL TRIAL: NCT05757726
Title: Feasibility Study of the Velocity™ Percutaneous Arterio-Venous Fistula System
Brief Title: Early Feasibility of the Velocity™ Percutaneous PAVF System
Acronym: VENOS-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venova Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CP0251.A
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-10

CONDITIONS: Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Interventional Arm (Experimental)
  Interventions: Device: Velocity pAVF system

INTERVENTIONS:
Device: Velocity pAVF system — A second generation percutaneous AVF device that creates an AVF between the proximal radial artery and cubital perforating vein.

SUMMARY:
An early feasibility study of the the initial safety and efficacy of the Velocity Percutaneous Arterio-Venous Fistula (pAVF) System when used to percutaneously create an arteriovenous fistula in patients with ESRD requiring hemodialysis vascular access.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosed with ESRD and currently on hemodialysis for less than 12 months using a central venous catheter for access
* Eligible for a native surgical brachiocephalic arteriovenous fistula following assessment by the principal investigator and study sponsor
* Cubital perforating vein diameter of > 2.5 mm and length > 10.0 mm
* Proximal radial artery diameter ≥ 2.0 mm
* Patient is free of clinically significant conditions or illness within 30 days prior to the AV fistula that may compromise the procedure
* Willing and competent to give written informed consent

Exclusion Criteria:

* Distance between Proximal Radial Artery and Cubital Perforating vein > 3mm
* Ipsilateral arm systolic blood pressure < 110 mmHg
* Known central venous stenosis or central vein narrowing > 50% ipsilateral to the study extremity
* Any obstruction of venous outflow from device implant site to the axillary vein
* Patients with occlusion of the ulnar or radial artery at any level or an abnormal Allen's test
* Any previous dialysis vascular access procedures in the study extremity
* History of steal syndrome (hand ischemia) from a previous hemodialysis vascular access of the non-study extremity which required intervention or access abandonment
* Upper extremity venous occlusion(s) and/or vessel abnormality(ies) of the study extremity that precludes endovascular AVF creation as determined by principal investigator or study sponsor
* Evidence of active systemic infections on day of the procedure or infection at the access site within the past 7 days
* History or evidence of severe cardiac disease (NYHA Functional Class III or IV), myocardial infarction within six months prior to study entry, ventricular tachyarrhythmias requiring continuing treatment, or unstable angina
* Currently being treated with another investigational device or drug
* Known adverse effects to sedation and/or anesthesia which cannot be adequately pre-medicated
* Uncontrolled or poorly controlled diabetes defined as a HbA1C > 10%
* Hypercoagulable condition, bleeding diathesis or coagulation disorder
* Receiving anti-coagulant therapy that cannot be safely held in the peri-procedural period
* Edema of the upper arm of the study extremity
* Scheduled kidney transplant within 6 months of enrollment
* Peripheral white blood cell count < 1.5 K/mm3 or platelet count < 75,000 cells/mm3
* Current diagnosis of carcinoma (defined as in remission < 1 year)
* Pregnant or currently breast feeding
* History of substance abuse or anticipated to be non- compliant with medical care or study requirements based on investigator judgment
* Allergies to NiTi alloy or any of the components of the Velocity Implant or Delivery System
* Written informed consent not obtainable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Procedural Success | Immediate
  Defined as Velocity deployment and delivery system withdrawal with intraprocedural duplex ultrasound demonstrating arterialized flow in the cephalic vein 2 cm central from the pAVF anastomosis
Serious Adverse Device Events | 6 weeks
  Defined as any Serious Adverse Event that reasonably suggests is caused by the device or procedure.
Major Reintervention | 6 weeks
  Defined as any open surgery, thrombectomy or thrombolysis in the index limb following pAVF creation.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Ebner, MD, Principal Investigator — Sanatorio Italiano
Locations (1):
- Sanatorio Italiano, Asunción, Paraguay